CLINICAL TRIAL: NCT03042156
Title: Immunotherapy And Palliative Radiotherapy Combined In Patients With Advanced Malignancy
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 16-6189
Record Dates: First submitted 2016-12-28; First posted 2017-02-03 (Estimated); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Palliative; Advanced Cancer; Immunotherapy; Radiation Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: Palliative Radiation Therapy

SUMMARY:
Immunotherapy includes a class of medication called checkpoint inhibitors, which are a relatively new medication therapy for many types of cancer which are metastatic, meaning it has spread to other parts of the body.Immune therapy medication may be given safely with radiation treatment, and in rare cases it may even make radiotherapy more effective. When radiation therapy is given in the "palliative" setting it is given to treat pain/discomfort and not necessarily shrink or get rid of the tumour. Palliative radiotherapy may be given for many reasons, but common examples include painful bone or liver tumours, brain metastases, or symptoms from a chest tumour such as feeling breathless, cough, or bleeding. Palliative radiotherapy is usually given in smaller amounts and less frequently than other types of radiation therapy. Because checkpoint inhibitors are relatively new there is not a huge amount of evidence looking at how patients respond when the treatments are combined, or in which patients immune therapy may make radiation therapy even more effective. This study is looking at the way patients who are on or about to start immune therapy and who have been recommended for palliative radiotherapy, respond to the combination of these two treatments.

The purpose of this study is to describe the treatment outcomes in patients with cancer that has spread who are managed with a combination of immune therapy medication and radiotherapy. This research is being done because there is limited information about the outcomes of combined immune therapy and radiotherapy treatment from a patient's perspective, but also in terms of which patients may have a better response to combined treatment. In particular, the study aims to describe how combined treatment affects cancer not only in the area where radiotherapy is given, but also outside the part of the body that receives radiotherapy (which is called "abscopal" effect).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years or older
2. Histologically or cytologically confirmed solid tumor malignancy
3. Advanced disease (locally advanced and/or metastatic)
4. Life expectancy > 3 months
5. Patients planned to receive palliative radiotherapy (including whole liver radiotherapy)
6. Patients who are already on or about to commence a checkpoint inhibitor
7. Measurable disease according to irRECIST on CT or MRI
8. ECOG performance status 0-2
9. Able to provide informed consent
10. Able to complete telephone/email communication
11. Additional criteria for subset of patients for abscopal analysis (to be done post hoc):

    1. Measurable disease outside irradiated volume
    2. Must be on same checkpoint inhibitor/immunotherapy (or same class of checkpoint inhibitor) for 3 months prior to radiotherapy and have stable disease or oligoprogression in past 3 months
    3. Availability of prior biopsy specimen (preferably fresh frozen tissue) for research and genotyping

Exclusion Criteria:

1. Medical conditions which may be contraindications to radiotherapy
2. Any medical or non-medical issue that would affect the patient's ability to provide informed consent for study participation, or would interfere with the patient's treatment on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced malignancy referred for palliative radiotherapy for symptom control who are either (a) already on a checkpoint inhibitor or (b) about to start immunotherapy (including PD1 inhibitors, CTLA4 inhibitors or other novel checkpoint inhibitor agents)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of patients showing rates of grade 3 or higher toxicity | 4 months
  Toxicity and safety data for combined therapy with immunotherapy and palliative RT (documentation that the rates of grade 3 or higher toxicity with combined therapy is < 30%) using patient reported outcomes (symptoms, toxicities, quality of life measures), clinical outcomes (physical examination, and CT imaging results) at baseline, 1 and 3 months post radiotherapy.
  Only the highest toxicity/per patient will be used for analysis, regardless of the time point of when the information is collected

SECONDARY OUTCOMES:
In-field response on imaging and evidence of out of field (abscopal) response. | 4 months
  Documentation of efficacy using CT imaging at 1 and 3 months post radiotherapy.
The number of ESAS questionnaires completed with the aid of a caregiver | 1 year
  Gather information on the efficacy collecting PRO's via in person or phone using questionnaires
biomarkers analyses as an indicator of abscopal response | 4 months
  Optional for consenting patients, done at 1 and 3 months post radiotherapy.
The number of EQ5D questionnaires completed with the aid of a caregive | 1 year
  Gather information on the efficacy collecting PRO's via in person or phone using questionnaires

OTHER OUTCOMES:
inflammatory and radiation sensitivity signatures from genotyping using archival tissue | 1 year
  Optional - from consenting patients (n=10) who already have readily available archival tumour tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada